CLINICAL TRIAL: NCT00997113
Title: Physiologic Stress During Procedural Sedation With and Without Alfentanil
Brief Title: Stress During Deep Sedation With Propofol With and Without Alfentanil
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hennepin Healthcare Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MMRF093051
Record Dates: First submitted 2009-10-12; First posted 2009-10-19 (Estimated); Results first posted 2014-09-25 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Sedation
Keywords: propofol; alfentanil; procedural sedation; stress biomarkers; Deep procedural sedation in the ED
MeSH Terms: interventions — Propofol; Alfentanil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Propofol (Active Comparator): propofol only for deep procedural sedation
  Interventions: Drug: propofol
- Propofol/alfentanil (Active Comparator): Propofol with alfentanil for deep procedural sedation
  Interventions: Drug: propofol; Drug: alfentanil

INTERVENTIONS:
Drug: propofol — 1 mg/kg IV followed by 0.5 mg/kg iv prn sedation
Drug: alfentanil — alfentanil 10 ug/kg immediately prior to propofol dose
  Arms: Propofol/alfentanil

SUMMARY:
This is a randomized clinical trial of deep procedural sedation with propofol with and without supplemental alfentanil. Patients will be assessed for total and fractionated serum catecholamines before and after the procedure in addition to usual procedural sedation outcomes parameters to assess the adrenergic effect of propofol sedation without supplemental opioid.

ELIGIBILITY:
Inclusion Criteria:

* patients who will require deep procedural sedation with propofol in the ED

Exclusion Criteria:

* age <18
* intoxication
* unable to provide informed consent
* allergy to propofol or alfentanil
* pregnant
* ASA physical status score > 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-10; Primary Completion 2012-10 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James R. Miner, MD, Principal Investigator — Hennepin Faculty Associates
Locations (1):
- Hennepin County Medical Center, Minneapolis, Minnesota, United States

REFERENCES:
- [Result] Miner JR, Moore JC, Plummer D, Gray RO, Patel S, Ho JD. Randomized clinical trial of the effect of supplemental opioids in procedural sedation with propofol on serum catecholamines. Acad Emerg Med. 2013 Apr;20(4):330-7. doi: 10.1111/acem.12110. PMID 23701339

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 34 patients were elligible, 14 underwent sedation emergently before the patient could be approached for study enrollment.
Period: Overall Study
Arm/Group | Propofol | Propofol/Alfentanil
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Propofol | Propofol/Alfentanil | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Median (Full Range); unit: years] | 34 [18 to 60] | 36 [20 to 58] | 35 [18 to 60]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 6 | 4 | 10
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in Serum Catecholamines
Description: change in serum catecholamine levels, values indicate a decrease over the procedure. These patients underwent fracture reduction procedures which are typically associated with an increase in catecholamines.
Time Frame: one minute prior to the start of the procedure and immediately at the end of sedation procedure (median time of procedure 12 minutes range 6-26 minutes
Measure: Median (Inter-Quartile Range); unit: mcg/ml
Arm/Group | Propofol | Propofol/Alfentanil
Number analyzed (Participants) | 10 | 10
mcg/ml | 87 [1 to 353] | 106 [21 to 295]
Statistical Analysis 1: Comparison: Propofol vs Propofol/Alfentanil; Comparison of the change in serum catecholamines from one minute before the procedure to one minute after. In order to detect a 20% difference in mean catecholamine values between groups, assuming a 30% standard deviation, with an alpha of 0.05 and a beta of 0.2 (80% power), power analysis indicated that 10 patients per group were required; Test type: Superiority or Other; p = 0.940, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Respiratory Depression
Description: categorized as a change in end tidal CO2 from baseline >10mmhg, a loss of end tidal CO2 waveform for more than 6 seconds, or an oxygen saturation less than 93%.
Time Frame: From one minute prior to the start of the sedation procedure until the patient has returned to baseline mental status
Measure: Number; unit: participants
Arm/Group | Propofol | Propofol/Alfentanil
Number analyzed (Participants) | 10 | 10
participants | 4 | 5

3. Secondary Outcome: Patient Reported Pain and Recall of the Painful Procedure for Which They Were Sedated Measure by Patient Query After They Had Regained Their Baseline Level of Consciousness After the Procedure
Description: Pain and recall were measured seperately by direct patient query. The patient was asked if they experienced any pain during the procedure. The patient was then asked if they could recall any part of the fracture reduction. Patients who had either pain with the procedure of recall of the procedure were counted as having pain or recall with the procedure.
Time Frame: single time point measured after sedation procedure completed
Measure: Number; unit: participants
Arm/Group | Propofol | Propofol/Alfentanil
Number analyzed (Participants) | 10 | 10
participants | 2 | 5

ADVERSE EVENTS:
Arm/Group | Propofol | Propofol/Alfentanil
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 1/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Propofol (N=10) | Propofol/Alfentanil (N=10)
apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — patient inadvertently given 5 times the study dose of alfentanil, developed apnea that resovled with bag valve mask ventilation over 2 minutes, resolved completely after 2 minutes without subsequent difficulty

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No